CLINICAL TRIAL: NCT02420288
Title: Effect of Physical Exercise Program on Fetoplacental Growth: a Randomized Controlled Trial
Brief Title: Effect of Physical Exercise Program on Fetoplacental Growth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Marina Vargas Terrones, PhD student, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INEF-001
Record Dates: First submitted 2015-04-08; First posted 2015-04-17 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Pregnancy; Healthy
Keywords: Pregnancy; Fetoplacental growth; Physical exercise; Pregnant; Placental development; Active pregnancy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Pregnant women not participating in supervised physical exercise program. The subjects in this group will be monitored during pregnancy to know if they make any kind of exercise on your own, to know which are really sedentary pregnant women.
- Exercise Group (Experimental): Pregnant women participating in supervised physical exercise program.
  Interventions: Behavioral: Exercise Group

INTERVENTIONS:
Behavioral: Exercise Group — Supervised physical conditioning program of three 55-60 minute sessions per week during whole pregnancy (before week 16 to 38). Each session consists of 25-30 minutes of cardiovascular exercise,10 minutes of specific exercises (strength and balance exercises), and 10 minutes of pelvic floor muscles training.
  Aerobic activity was prescribed at light to moderate intensity, aiming for 55-60% of heart rate reserve. All subjects wore a heart rate (HR) monitor (Polar FT7) during the training sessions to ensure that exercise intensity was light to moderate.
  Other Names: Supervised physical exercise program group
  Arms: Exercise Group

SUMMARY:
The aim of this study is to examine the effect of a supervised physical exercise program during pregnancy on fetoplacental growth.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines
* Being able to communicate in spanish
* Giving birth at Hospital Universitario de Torrejón, Hospital Universitario de Puerta de Hierro or Hospital Universitario Severo Ochoa (Madrid)

Exclusion Criteria:

* Multiparity
* Obstetrician complications
* Being interested in the study after 18 weeks
* Not having availability to attend to the physical exercise program
* Younger than 18 years old
* Older than 45 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Placental weight | At delivery
Fetal birth weight | At delivery
Change from baseline in maternal gestational weight | 38-42 weeks of gestation
  Maternal weight gain during pregnancy. Weight will be measured at the beginning and at the end of the pregnancy

SECONDARY OUTCOMES:
Pregestational weight and Body Mass Index (BMI) | Before pregnancy
pH umbilical cord | At delivery
Fetal size outcomes | At delivery
  Size and height, head circumference and body mass index of the baby
Fetal glycemia level | At delivery
Apgar score | At delivery
  Apgar score will be valued 1 and 5 minutes after delivery
Maternal delivery outcomes (composite) | At delivery
  Type of labor, stage and duration of labor
Postpartum depression | 0-12 postpartum months
  The level of maternal depression after delivery will be measured with the Edinburgh Postnatal Depression Scale (EPDS)
Changes from baseline in prenatal depression | Up to 36 weeks
  The level of maternal depression during pregnancy will be measured at the beginning and at the end of the pregnancy, as well as at 8 weeks postpartum, with the Center for Epidemiologic Studies Depression Scale (CES-D)
Changes from baseline in maternal quality of life | Up to 36 weeks
  Maternal quality of life will be measured at the beginning and at the end of the pregnancy, as well as at 8 weeks postpartum, with the Short Form-36 Health Survey (SF-36)
Changes from baseline in urinary incontinence | Up to 36 weeks
  Urinary incontinence will be measured at the beginning and at the end of the pregnancy, as well as at 8 weeks postpartum, with the International Consultation on Incontinence Questionnaire Short-Form (ICIQ-SF)
Gestational diabetes | 24-28 weeks
  Gestational diabetes will be measured with the O' Sullivan's test

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Barakat Carballo, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Spain

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Vargas-Terrones M, Barakat R, Santacruz B, Fernandez-Buhigas I, Mottola MF. Physical exercise programme during pregnancy decreases perinatal depression risk: a randomised controlled trial. Br J Sports Med. 2019 Mar;53(6):348-353. doi: 10.1136/bjsports-2017-098926. Epub 2018 Jun 13. PMID 29899050
- [Derived] Barakat R, Vargas M, Brik M, Fernandez I, Gil J, Coteron J, Santacruz B. Does Exercise During Pregnancy Affect Placental Weight?: A Randomized Clinical Trial. Eval Health Prof. 2018 Sep;41(3):400-414. doi: 10.1177/0163278717706235. Epub 2017 Apr 25. PMID 29179559
- See also: Website that provides information about our research group projects — http://afipe.es/embarazo-y-ejercicio.html